CLINICAL TRIAL: NCT02551042
Title: A Phase II, Double-blind, Randomized, Placebo-controlled Study to Investigate Pharmacokinetics (PK), Safety and Efficacy of Intravenous Factor XIII Treatment in Patients With Systemic Sclerosis
Brief Title: CSL Behring Sclero XIII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13/0417; 2014-001101-40 (EudraCT Number)
Record Dates: First submitted 2014-12-17; First posted 2015-09-16 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Systemic Sclerosis
Keywords: Digital Ulcers; Raynauds Phenomenon; Factor XIII
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers; Raynaud Disease | interventions — Factor VIII; Factor XIII; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment arm (Experimental): Fibrogammin®P, coagulation factor XIII concentrate (Human) IV infusion
  Interventions: Drug: Fibrogammin®P, coagulation factor XIII concentrate (Human)
- Placebo arm (Placebo Comparator): Placebo will be 0.9 % Sodium chloride solution IV infusion
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Fibrogammin®P, coagulation factor XIII concentrate (Human) — IV infusion
  Other Names: Factor XIII
  Arms: Active treatment arm
Drug: 0.9% sodium chloride — IV infusion
  Other Names: Normal saline
  Arms: Placebo arm

SUMMARY:
Many patients with Scleroderma (Systemic sclerosis) experience damage to blood vessels, mainly to the small arteries. A common manifestation of this is Raynaud's phenomenon (fingers or toes turning white then blue in the cold) and digital ulcers (open sores on the fingertips). The purpose of this study is to see how effective the study drug Human Factor XIII Concentrate is in treating patients who have these and other common manifestation of Scleroderma. It will be given in addition to the accepted treatments used for this disease.

DETAILED DESCRIPTION:
This is a phase II, double-blind, randomized, placebo-controlled study to investigate pharmacokinetics (PK), safety and efficacy of intravenous factor XIII treatment in patients with systemic sclerosis.

Scleroderma (Systemic sclerosis) is a multisystem rheumatic disease that is characterised by progressive vascular damage e.g Raynaud's phenomenon and digital ulcers and organ fibrosis e.g. skin thickening and pulmonary fibrosis.The disease is associated with significant morbidity and mortality and current therapeutic options are only partially effective, including Cyclophosphamide for skin or lung fibrosis and Bosentan which reduces but does not heal digital ulcers.

There is no cure available and there is therefore a high need for new therapeutic options.Administration of human Factor XIII (FXIII) concentrate in patients with scleroderma demonstrated promising results in the 1980s and 1990s . However these studies were not performed according to current Good Clinical Practice (GCP) guidelines and involved relatively small sample sizes.

This is a single site study, therefore all study participants will be seen at the Royal Free London National Health Service (NHS) Foundation Trust.Total study duration is 36 months and will involve 2 phases: an initial single dose, pharmacokinetic (PK) phase in 8 subjects over 6 weeks and a multiple dose, active treatment phase in 18 subjects over 24 weeks. During the treatment phase subjects will be randomized at 2:1 ratio to either FXIII or Placebo and will receive biweekly injection of either factor XIII Concentrate or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults.
* Subjects with a diagnosis of systemic sclerosis (scleroderma, SSc) according to the 2013 American College of Rheumatology European League Against Rheumatism (ACR EULAR) classification criteria. They will be classified according to LeRoy criteria as limited or diffuse subset.
* Females of childbearing potential must be willing to use a reliable form of medically acceptable contraception and have a negative pregnancy test.
* Subjects will have serological status for hepatitis A and B assessed at screening.
* Patients who have given their free and informed consent. -≥ 18 years.

Exclusion Criteria:

Participants must:

* Be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation (females of childbearing potential and males)
* Have a negative pregnancy test within 7 days prior to being registered for trial treatment (females of childbearing potential). NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Not be breastfeeding (females).

Participants must not:

* Have allergies to excipients of the investigational medicinal product (IMP) and placebo
* Have uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure ≥ 160 mmHg or sitting diastolic blood pressure ≥ 100 mmHg.
* Have portal hypertension or chronic liver disease defined as mild to severe hepatic impairment (Child-Pugh Class A-C). Subjects positive for Hepatitis C with evidence of active viral replication on sensitive polymerase chain reaction (PCR) testing are also excluded.
* Have hepatic dysfunction, defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≥ 3 times the upper limit of the normal range (× ULN) at the Screening Visit.
* Have chronic renal insufficiency as defined by a serum creatinine ≥ 2.5 mg/dL (≤ 221 micromol/L) or requires dialysis.
* Have a haemoglobin concentration ≤ 10 g/dL (≤ 100 g/L) at the Screening Visit.
* Have a history of left-sided heart disease and/or clinically significant cardiac disease, including but not limited to any of the following: aortic or mitral valve disease (stenosis or regurgitation) defined as more than minimum aortic insufficiency and more than moderate mitral regurgitation (stenosis or regurgitation≥ grade 1); pericardial constriction; restrictive or congestive cardiomyopathy; left ventricular ejection fraction ≤ 40 % by multiple gated acquisition scan (MUGA), angiography, or echocardiography; left ventricular shortening fraction ≤ 22 % by echocardiography; or symptomatic coronary disease with demonstrable ischemia.
* Have a history of malignancies within 5 years of Screening Visit with the exception of localized skin or cervical carcinomas.
* Have psychiatric, addictive, or other disorder that compromises the ability to give informed consent for participating in this study. This includes subjects with a recent history of abusing alcohol or illicit drugs.
* Be receiving ongoing treatment with hyperbaric oxygen
* Have pulmonary artery hypertension (PAH)
* Have received IV Iloprost within the last 2 months
* Have been treated with sympathectomy or toxin botulinum A within the last 3 months
* Have had thrombosis, stroke, pulmonary embolism or myocardial infarction in the last 6 months
* Have a diagnosis of diabetes mellitus requiring dietary restriction of carbohydrate.
* Be on a low sodium diet on medical advice.
* Be participating in another clinical trial involving an investigational medicinal product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome assessed by skin involvement measured with modified Rodnan skin score | 24 weeks
Primary outcome assessed by skin involvement measured with Raynaud condition score | 24 weeks

SECONDARY OUTCOMES:
Pulmonary function measured by pulmonary function test | 24 weeks
  Pulmonary function measured by pulmonary function test
Hand function measured with Cochin hand function | 24 weeks
  Hand function measured with Cochin hand function
Quality of life measured with Short Form-36 (SF-36) quality of life questionnaire | 24 weeks
  Quality of life measured with SF36 quality of life questionnaire
Number of new digital ulcers (DU) | 24 weeks
  Prevention of new DU: Number of new DU developed during a 24-week period of treatment
Complete healing of digital ulcers (DU) | 24 weeks
  Healing of DU: Complete healing of DUs present at baseline; each DU is considered as an entity
Digital ulcer pain assessment | 24 weeks
  DU Pain assessment at 4, 8, 12, 16, 24 weeks of treatment: Pain will be assessed by analogue scale for pain (Visual Analogue Scale, VAS)
Digital ulcer pain assessment | 24 weeks
  DU Pain assessment at 4, 8, 12, 16, 24 weeks of treatment: Pain will be assessed by Raynaud's severity (Raynaud's condition score)
Digital ulcer worsening: hospitalisation required | 24 weeks
  Number of overnight hospitalisations for digital ulcers
Digital ulcer worsening: surgical intervention required | 24 weeks
  Number of additional surgical treatments for digital ulcer in outpatient clinic
Digital ulcer worsening: Digital ulcer infection | 24 weeks
  Number of digital ulcers with infections
Digital ulcer worsening: Gangrene | 24 weeks
  Number of episodes of gangrene
Digital ulcer worsening: Amputation | 24 weeks
  Number of amputations
Digital ulcer worsening: Need of local sympathectomy | 24 weeks
  Number of local sympathectomies
Digital ulcer worsening: Need of toxin Botulinum A | 24 weeks
  Number of treatments with Botulinum toxin A
Digital ulcer worsening: Need of oral or parenteral antibiotic | 24 weeks
  Number of treatments needed with oral or parenteral antibiotic
Digital ulcer worsening: Need of intravenous (IV) Iloprost : this is considered treatment failure | 24 weeks
  Number of treatments needed with intravenous (IV) Iloprost : this is considered treatment failure

OTHER OUTCOMES:
Safety endpoints: Physical examination (including height, weight, BMI, digital ulcer characterization) | 24 weeks
  Physical examination (including height, weight, BMI, digital ulcer characterization)
Safety endpoints: Adverse events | 24 weeks
  Adverse events
Safety endpoints: Serious adverse events | 24 weeks
  Serious adverse events
Safety endpoints: ECG | 24 weeks
  ECG
Safety endpoints: Vital signs | 24 weeks
  Vital signs
Safety endpoints: Clinical laboratory parameters | 24 weeks
  Clinical laboratory parameters
Safety endpoints: Pregnancy | 24 weeks
  Serum or urine pregnancy tests will be performed at each visit and will be reported positive or negative
Safety endpoints -Adverse events of special interest: thromboembolic events | 24 weeks
  Adverse events of special interest: thromboembolic events

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Denton, PhD, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LeRoy EC, Black C, Fleischmajer R, Jablonska S, Krieg T, Medsger TA Jr, Rowell N, Wollheim F. Scleroderma (systemic sclerosis): classification, subsets and pathogenesis. J Rheumatol. 1988 Feb;15(2):202-5. No abstract available. PMID 3361530
- [Background] Nihtyanova SI, Brough GM, Black CM, Denton CP. Clinical burden of digital vasculopathy in limited and diffuse cutaneous systemic sclerosis. Ann Rheum Dis. 2008 Jan;67(1):120-3. doi: 10.1136/ard.2007.072686. Epub 2007 Jul 27. PMID 17660220
- [Background] Levy JH, Greenberg C. Biology of Factor XIII and clinical manifestations of Factor XIII deficiency. Transfusion. 2013 May;53(5):1120-31. doi: 10.1111/j.1537-2995.2012.03865.x. Epub 2012 Aug 28. PMID 22928875
- [Background] Yee VC, Pedersen LC, Le Trong I, Bishop PD, Stenkamp RE, Teller DC. Three-dimensional structure of a transglutaminase: human blood coagulation factor XIII. Proc Natl Acad Sci U S A. 1994 Jul 19;91(15):7296-300. doi: 10.1073/pnas.91.15.7296. PMID 7913750
- [Background] Nugent DJ. Prophylaxis in rare coagulation disorders -- factor XIII deficiency. Thromb Res. 2006;118 Suppl 1:S23-8. doi: 10.1016/j.thromres.2006.02.009. Epub 2006 Apr 17. PMID 16616323
- [Background] Ivaskevicius V, Seitz R, Kohler HP, Schroeder V, Muszbek L, Ariens RA, Seifried E, Oldenburg J; Study Group. International registry on factor XIII deficiency: a basis formed mostly on European data. Thromb Haemost. 2007 Jun;97(6):914-21. PMID 17549292
- [Background] Dallabrida SM, Falls LA, Farrell DH. Factor XIIIa supports microvascular endothelial cell adhesion and inhibits capillary tube formation in fibrin. Blood. 2000 Apr 15;95(8):2586-92. PMID 10753838
- [Background] Dardik R, Shenkman B, Tamarin I, Eskaraev R, Harsfalvi J, Varon D, Inbal A. Factor XIII mediates adhesion of platelets to endothelial cells through alpha(v)beta(3) and glycoprotein IIb/IIIa integrins. Thromb Res. 2002 Feb 15;105(4):317-23. doi: 10.1016/s0049-3848(02)00014-2. PMID 12031826
- [Background] Dardik R, Solomon A, Loscalzo J, Eskaraev R, Bialik A, Goldberg I, Schiby G, Inbal A. Novel proangiogenic effect of factor XIII associated with suppression of thrombospondin 1 expression. Arterioscler Thromb Vasc Biol. 2003 Aug 1;23(8):1472-7. doi: 10.1161/01.ATV.0000081636.25235.C6. Epub 2003 Jun 12. PMID 12805075
- [Background] Dardik R, Leor J, Skutelsky E, Castel D, Holbova R, Schiby G, Shaish A, Dickneite G, Loscalzo J, Inbal A. Evaluation of the pro-angiogenic effect of factor XIII in heterotopic mouse heart allografts and FXIII-deficient mice. Thromb Haemost. 2006 Mar;95(3):546-50. doi: 10.1160/TH05-06-0409. PMID 16525585
- [Background] Khanna D, Furst DE, Hays RD, Park GS, Wong WK, Seibold JR, Mayes MD, White B, Wigley FF, Weisman M, Barr W, Moreland L, Medsger TA Jr, Steen VD, Martin RW, Collier D, Weinstein A, Lally EV, Varga J, Weiner SR, Andrews B, Abeles M, Clements PJ. Minimally important difference in diffuse systemic sclerosis: results from the D-penicillamine study. Ann Rheum Dis. 2006 Oct;65(10):1325-9. doi: 10.1136/ard.2005.050187. Epub 2006 Mar 15. PMID 16540546
- [Background] Kilian O, Fuhrmann R, Alt V, Noll T, Coskun S, Dingeldein E, Schnettler R, Franke RP. Plasma transglutaminase factor XIII induces microvessel ingrowth into biodegradable hydroxyapatite implants in rats. Biomaterials. 2005 May;26(14):1819-27. doi: 10.1016/j.biomaterials.2004.06.015. PMID 15576156
- [Background] Mirochnik Y, Kwiatek A, Volpert OV. Thrombospondin and apoptosis: molecular mechanisms and use for design of complementation treatments. Curr Drug Targets. 2008 Oct;9(10):851-62. doi: 10.2174/138945008785909347. PMID 18855619
- [Background] Nor JE, Mitra RS, Sutorik MM, Mooney DJ, Castle VP, Polverini PJ. Thrombospondin-1 induces endothelial cell apoptosis and inhibits angiogenesis by activating the caspase death pathway. J Vasc Res. 2000 May-Jun;37(3):209-18. doi: 10.1159/000025733. PMID 10859480
- [Background] Streit M, Velasco P, Riccardi L, Spencer L, Brown LF, Janes L, Lange-Asschenfeldt B, Yano K, Hawighorst T, Iruela-Arispe L, Detmar M. Thrombospondin-1 suppresses wound healing and granulation tissue formation in the skin of transgenic mice. EMBO J. 2000 Jul 3;19(13):3272-82. doi: 10.1093/emboj/19.13.3272. PMID 10880440
- [Background] Dardik R, Loscalzo J, Eskaraev R, Inbal A. Molecular mechanisms underlying the proangiogenic effect of factor XIII. Arterioscler Thromb Vasc Biol. 2005 Mar;25(3):526-32. doi: 10.1161/01.ATV.0000154137.21230.80. Epub 2004 Dec 23. PMID 15618543
- [Background] Dardik R, Loscalzo J, Inbal A. Factor XIII (FXIII) and angiogenesis. J Thromb Haemost. 2006 Jan;4(1):19-25. doi: 10.1111/j.1538-7836.2005.01473.x. Epub 2005 Aug 26. PMID 16129024
- [Background] Gabrielli A, Avvedimento EV, Krieg T. Scleroderma. N Engl J Med. 2009 May 7;360(19):1989-2003. doi: 10.1056/NEJMra0806188. No abstract available. PMID 19420368
- [Background] Macko RF, Gelber AC, Young BA, Lowitt MH, White B, Wigley FM, Goldblum SE. Increased circulating concentrations of the counteradhesive proteins SPARC and thrombospondin-1 in systemic sclerosis (scleroderma). Relationship to platelet and endothelial cell activation. J Rheumatol. 2002 Dec;29(12):2565-70. PMID 12465153
- [Background] Mimura Y, Ihn H, Jinnin M, Asano Y, Yamane K, Tamaki K. Constitutive thrombospondin-1 overexpression contributes to autocrine transforming growth factor-beta signaling in cultured scleroderma fibroblasts. Am J Pathol. 2005 May;166(5):1451-63. doi: 10.1016/s0002-9440(10)62362-0. PMID 15855645
- [Background] Avouac J, Clemessy M, Distler JH, Gasc JM, Ruiz B, Vacher-Lavenu MC, Wipff J, Kahan A, Boileau C, Corvol P, Allanore Y. Enhanced expression of ephrins and thrombospondins in the dermis of patients with early diffuse systemic sclerosis: potential contribution to perturbed angiogenesis and fibrosis. Rheumatology (Oxford). 2011 Aug;50(8):1494-504. doi: 10.1093/rheumatology/keq448. Epub 2011 Mar 30. PMID 21454305
- [Background] Farina G, Lafyatis D, Lemaire R, Lafyatis R. A four-gene biomarker predicts skin disease in patients with diffuse cutaneous systemic sclerosis. Arthritis Rheum. 2010 Feb;62(2):580-8. doi: 10.1002/art.27220. PMID 20112379
- [Background] Paye M, Nusgens BV, Lapiere CM. Factor XIII of blood coagulation modulates collagen biosynthesis by fibroblasts in vitro. Haemostasis. 1989;19(5):274-83. doi: 10.1159/000215988. PMID 2777140
- [Background] Denton CP, Zheng B, Evans LA, Shi-wen X, Ong VH, Fisher I, Lazaridis K, Abraham DJ, Black CM, de Crombrugghe B. Fibroblast-specific expression of a kinase-deficient type II transforming growth factor beta (TGFbeta) receptor leads to paradoxical activation of TGFbeta signaling pathways with fibrosis in transgenic mice. J Biol Chem. 2003 Jul 4;278(27):25109-19. doi: 10.1074/jbc.M300636200. Epub 2003 Apr 21. PMID 12707256
- [Background] Crawford SE, Stellmach V, Murphy-Ullrich JE, Ribeiro SM, Lawler J, Hynes RO, Boivin GP, Bouck N. Thrombospondin-1 is a major activator of TGF-beta1 in vivo. Cell. 1998 Jun 26;93(7):1159-70. doi: 10.1016/s0092-8674(00)81460-9. PMID 9657149
- [Background] Thivolet J, Perrot H, Meunier F, Bouchet B. [Therapeutic action of coagulation factor XIII in scleroderma. 20 cases]. Nouv Presse Med. 1975 Nov 15;4(39):2779-82. French. PMID 1105424
- [Background] Delbarre F, Godeau P, Thivolet J. Factor XIII treatment for scleroderma. Lancet. 1981 Jul 25;2(8239):204. doi: 10.1016/s0140-6736(81)90385-8. No abstract available. PMID 6114269
- [Background] Guillevin L, Chouvet B, Mery C, Thivolet J, Godeau P, Delbarre F. [Treatment of generalized scleroderma with factor XIII. Study of 25 cases]. Rev Med Interne. 1982;3(3):273-7. doi: 10.1016/s0248-8663(82)80031-3. No abstract available. French. PMID 6758093
- [Background] Guillevin L, Euller-Ziegler L, Chouvet B, De Gery A, Chassoux G, Lafay P, Ziegler G, Godeau P, Amor B, Thivolet J. [Treatment of systemic scleroderma with factor XIII in 86 patients, with long-term follow-up]. Presse Med. 1985 Dec 28;14(46):2327-9. French. PMID 2935830
- [Background] Euller-Ziegler L, Corolleur YR, Marcou J, Commandre F, Grisot C, Ziegler G. [Long-term treatment of systemic scleroderma with coagulation factor XIII. Developmental monitoring, especially of respiratory function]. Rev Rhum Mal Osteoartic. 1984 Oct;51(9):503-5. No abstract available. French. PMID 6505601
- [Background] Maekawa Y, Nogita T, Yamada M. Favorable effects of plasma factor XIII on lower esophageal sphincter pressure of progressive systemic sclerosis. Arch Dermatol. 1987 Nov;123(11):1440-1. No abstract available. PMID 3674907
- [Background] Guillevin L, Chouvet B, Mery C, De Gery A, Thivolet J, Godeau P, Delbarre F. Treatment of progressive systemic sclerosis using factor XIII. Pharmatherapeutica. 1985;4(2):76-80. PMID 3903781
- [Background] Quillinan NP, McIntosh D, Vernes J, Haq S, Denton CP. Treatment of diffuse systemic sclerosis with hyperimmune caprine serum (AIMSPRO): a phase II double-blind placebo-controlled trial. Ann Rheum Dis. 2014 Jan;73(1):56-61. doi: 10.1136/annrheumdis-2013-203674. Epub 2013 Sep 25. PMID 24067785
- See also: NovoThirteen® Summary of Product Characteristics — http://ec.europa.eu/health/documents/community-register/2012/20120903123586/anx_123586_en.pdf